CLINICAL TRIAL: NCT06618534
Title: Effectiveness of Azithromycin in Eradicating Nasopharyngeal Carriage of N. Meningitidis
Brief Title: Azithromycin for Meningococcal Carriage
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Georgia Department of Public Health (Unknown)
Responsible Party: Principal Investigator, Paulina Rebolledo, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008433; CDC-STUDY00008433 (Other: Centers for Disease Control and Prevention); 2025P012505 (Other: Emory IRB)
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Meningococcal Infections
MeSH Terms: conditions — Meningococcal Infections | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Azithromycin (Experimental): Persons with microbiologic documentation of N. meningitidis carriage will receive a single, standard dose of azithromycin.
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — A standard dose of azithromycin (500 mg) will be delivered by oral route.

SUMMARY:
The purpose of this study is to determine the effectiveness of azithromycin in the eradication of nasopharyngeal carriage of N. meningitidis

DETAILED DESCRIPTION:
Azithromycin belongs to the class of antimicrobials known as macrolides. They are approved for the treatment of a wide variety of infections, including community-acquired respiratory tract infections and sexually transmitted infections caused by different bacteria. Their mechanism of action is dependent on bacterial ribosomal binding, leading to inhibition of bacterial protein synthesis. Azithromycin has a broad spectrum of activity to include Gram-positive and Gram-negative organisms, as well as atypical and mycobacterial organisms.

A single oral dose of 500mg of azithromycin has been shown to eradicate N. meningitidis colonization. Historically, azithromycin has not been recommended as first-line chemoprophylaxis for close contacts of patients with invasive meningococcal disease (IMD) since it has not been well studied for this indication. A study from 2020 evaluated the activity of azithromycin against 205 invasive N. meningitidis isolates and found that 100% were susceptible according to Clinical and Laboratory Standards Institute (CLSI) breakpoints. Moreover, with the rise in cases of meningococcal disease caused by ciprofloxacin-resistant strains, the Centers for Disease Control and Prevention (CDC) recently updated their guidance to health department for when to consider other options (including azithromycin).

Participants identified as carriers of N. meningitidis will be asked to take a one-time oral dose of azithromycin, 500mg (standard dose).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide their own informed consent and understand study procedures
* Undergraduate and graduate students attending Emory University affiliated campuses who reside in university affiliated housing (for undergraduate/graduate) or in off-campus housing (undergraduates).

Exclusion Criteria:

* University faculty and staff
* Currently pregnant or breast feeding
* History of immediate or moderate-to-severe allergic reactions to azithromycin
* Individuals who have taken systemic antibiotics for any reason in the 30 days prior to enrollment
* Individuals with any symptoms of acute illness at the time of screening

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1120 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Eradication of N. meningitidis carriage | Day 7 (immediately prior to azithromycin administration), Day 21 (2 weeks after azithromycin administration)
  Eradication of N. meningitidis carriage is defined as positive culture at the second visit (immediately prior to azithromycin administration) and negative culture approximately 2 weeks after antibiotic administration.

SECONDARY OUTCOMES:
Proportion of Participants Culture-Positive | Day 1 (screening visit)
  Carriage prevalence is examined as the proportion of participants who are culture-positive at the initial visit, by serogroup and meningococcal vaccination status.
Minimal Inhibitory Concentrations (MICs) for Ciprofloxacin | Day 7 (immediately prior to azithromycin administration), Day 21 (2 weeks after azithromycin administration)
  The minimum inhibitory concentrations (MICs) are the lowest concentration of an antimicrobial that will inhibit the visible growth of a microorganism following overnight incubation. The MICs for ciprofloxacin among meningococcal isolates before and after azithromycin administration will be examined.
Minimal Inhibitory Concentrations (MICs) for Rifampin | Day 7 (immediately prior to azithromycin administration), Day 21 (2 weeks after azithromycin administration)
  The minimum inhibitory concentrations (MICs) are the lowest concentration of an antimicrobial that will inhibit the visible growth of a microorganism following overnight incubation. The MICs for rifampin among meningococcal isolates before and after azithromycin administration will be examined.
Minimal Inhibitory Concentrations (MICs) for Ceftriaxone | Day 7 (immediately prior to azithromycin administration), Day 21 (2 weeks after azithromycin administration)
  The minimum inhibitory concentrations (MICs) are the lowest concentration of an antimicrobial that will inhibit the visible growth of a microorganism following overnight incubation. The MICs for ceftriaxone among meningococcal isolates before and after azithromycin administration will be examined.
Minimal Inhibitory Concentrations (MICs) for Azithromycin | Day 7 (immediately prior to azithromycin administration), Day 21 (2 weeks after azithromycin administration)
  The minimum inhibitory concentrations (MICs) are the lowest concentration of an antimicrobial that will inhibit the visible growth of a microorganism following overnight incubation. The MICs for azithromycin among meningococcal isolates before and after azithromycin administration will be examined.
Risk Factors for Meningococcal Carriage | Day 1 (screening visit)
  Risk factors contributing to meningococcal carriage will be assessed by administering a survey to participants asking about their meningococcal vaccination status, recent antibiotic use, recent respiratory illness, smoke exposure and other social behaviors, with responses given in a "yes" or "no" format.

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Rebolledo, MD, MSc, Principal Investigator — Emory University
Locations (1):
- Hope Clinic of the Emory Vaccine Center, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Bacterial genome sequences will be deposited in "Public databases for molecular typing and microbial genome diversity" (PubMLST).
Supporting Information: Study Protocol
Time Frame: Individual participant data will be available for sharing following publication of results from this study, with no end date.
Access Criteria: Data will be made available for sharing with anyone who wishes to access the data, for any purpose. Data will be accessed via https://pubmlst.org/